CLINICAL TRIAL: NCT06888895
Title: Comparison of the Immediate Effect of Passive vs. Passive-Active Hamstring Stretching on Flexibility in Patients With Chronic Low Back Pain: Protocol for a Randomized Controlled Trial: EFIM2
Brief Title: Comparison of the Immediate Effect of Passive vs. Passive-Active Hamstring Stretching on Flexibility in Patients With Chronic Low Back Pain
Acronym: EFIM2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RBHP 2024 DOBIJA; 2024-A02351-46 (Other: ANSM)
Record Dates: First submitted 2025-03-06; First posted 2025-03-21 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: hamstring; chronic low back pain; extensibility deficit; passive stretching
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The same investigator will conduct both pre- and post-intervention assessments but will not be involved in administering the intervention for any patient, ensuring they remain blinded to patient allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive stretching (PS) (Active Comparator): In the control group, participants will receive one minute of passive hamstring stretching applied three times for each lower limb, with a 30-second rest time between stretches. This ensures that the intervention time is consistent across both groups, totaling approximately 15-20 minutes.
  Interventions: Other: Passive hamstring stretching
- Passive-Active Stretching (PAS) (Experimental): The passive-active stretching (PAS) intervention has two phases. In the first, a physiotherapist performs bilateral passive hamstring stretching, followed by a 30-second walk. The second phase includes three exercises with 30-second rest intervals between them.
  Active Knee Extension: The participant lies on their back with one thigh vertical (hip at 90°). A Stabilizer® Pressure Bio-feedback device is placed behind the lumbar spine to help maintain neutral position. The participant maintains 40 mmHg pressure while extending the knee to its maximum. Ten repetitions with a 3-second hold are performed.
  One-Leg Deadlift: While balancing on one leg, the participant bends forward and lifts the opposite leg, targeting hamstring elongation. Ten repetitions with a 5-second hold are performed.
  Bear-Squat Exercise: Starting in all-fours, participants shift weight onto toes and hands, moving the pelvis backward to elongate the hamstrings. Ten repetitions are performed.
  Interventions: Other: Passive-active stretching (PAS)

INTERVENTIONS:
Other: Passive-active stretching (PAS) — Passive-active stretching (PAS) combines conventional passive stretching with active exercises designed to activate muscles that promote hamstring elongation. On the other hand, passive stretching (PS) is a commonly administered intervention to improve hamstring flexibility.
  Other Names: Passive stretching (PS)
  Arms: Passive-Active Stretching (PAS)
Other: Passive hamstring stretching — Participants will receive one minute of passive hamstring stretching applied three times for each lower limb, with a 30-second rest time between stretches.
  Arms: Passive stretching (PS)

SUMMARY:
The goal of this clinical trial is to determine whether a combination of passive and active hamstring stretching (PAS) is more effective than passive stretching alone (PS) in improving flexibility in patients with chronic low back pain (CLBP).

The main questions it aims to answer are:

Does PAS lead to greater improvements in active flexibility compared to PS? Does PAS provide additional benefits in passive flexibility, hamstring stiffness, and pelvic tilt? Researchers will compare the PAS group and the PS group to see if combining passive and active stretching results in greater improvements in flexibility and movement control.

Participants will:

Perform either PAS or PS stretching exercises as assigned. Undergo measurements of flexibility, hamstring stiffness, and pelvic tilt before and after the intervention.

Answer a question about their perceived change in flexibility following the intervention.

This study aims to improve rehabilitation strategies for people with CLBP, helping them achieve better movement and pain relief.

DETAILED DESCRIPTION:
Individuals with chronic low back pain (CLBP) are affected by deficits in hamstring flexibility and lumbopelvic neuromuscular control. While passive hamstring stretching immediately improves passive hamstring flexibility, no clinically important difference in active range of motion has been observed.

The primary objective of the present randomized controlled study protocol is to compare the immediate effects of a novel combination of passive and active stretching (PAS) exercises with passive hamstring stretching (PS) alone on active flexibility.

The secondary objectives include conducting a similar comparison for passive flexibility, hamstring stiffness, and pelvic tilt, as well as estimating the Minimal Clinically Important Difference (MCID) for hamstring flexibility measures. Ninety CLBP patients will be randomized into PAS or PS group and will receive respective interventions. Primary outcome will be the mean value of two measurements of Active Knee Extension taken before and immediately after the intervention. Secondary outcomes, Fingertip-to-Floor distance, Straight Leg Raise, hamstring stiffness and pelvic tilt will be recorded and compared in the same manner. A group-by-time comparison will be conducted for primary and secondary outcomes. An anchor question about perceived by participants change in flexibility following intervention will serve to estimate MCID.

This study protocol is the first opportunity to assess whether combining passive and active hamstring stretching is better than passive stretching alone for achieving an immediate and clinically important improvement in active flexibility among CLBP patients. The results will provide valuable and time-efficient insights for the development of more comprehensive rehabilitation programs in both clinical and research settings.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 18 and 65 years
* Suffering from low-back pain for at least 3 months
* Presenting with hamstring flexibility deficit (Straight Leg Raise <85°, Fingertip-to-Floor distance >5 cm)

Exclusion Criteria:

* Patients with radicular pain
* Disc inflammation (MODIC Type 1)
* Other relevant pathologies (neurological, cardiovascular, respiratory, or oncological diseases)
* Significant surgical history (e.g., lumbar arthrodesis, knee or hip arthroplasty)
* Pregnancy or breastfeeding
* Patients under protective legal measures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Active Knee Extension (AKE) | Before and immediately after the intervention
  The Active Knee Extension (AKE) angle will be evaluated at baseline and immediately after the intervention. The mean value of the two measurements taken before the intervention will be compared with the mean value of two measurements taken immediately after the intervention. The change in AKE values of the less flexible lower limb, expressed as a percentage relative to the initial value, will be used to compare the effect between the PS and PAS groups.
  The participants will extend the tested knee as much as possible while keeping their thigh vertical against a plastic stick placed along the anterior surface of their thigh (maintaining 90° hip flexion). The rater will position the EasyAngle® digital inclinometer on the tibial crest, just below the tibial tuberosity, to record the maximal knee extension angle.

SECONDARY OUTCOMES:
Fingertip-to-Floor distance (FTF) | Before and immediately after the intervention
  The FTF distance will be evaluated at baseline and immediately after the intervention. The mean value of the two measurements taken before the intervention will be compared with the mean value of two measurements taken immediately after the intervention. The change in FTF values, expressed as a percentage relative to the initial value, will be used to compare the effect between the PS and PAS groups.
  The FTF measurement will be conducted in the standard manner by measuring the distance between the fingertips and the floor using a measuring tape at the end of the forward bending range, with knees fully extended.
Pelvic tilt angle | Before and immediately after intervention
  The pelvic tilt angle will be measured at baseline and immediately after the intervention. The mean value of the two measurements taken before the intervention will be compared with the mean value of two measurements taken immediately after the intervention. The change in pelvic tilt angle values, expressed as a percentage relative to the initial value, will be used to compare the effect between the PS and PAS groups.
  The EasyAngle® inclinometer will be placed on the sacrum to measure the sagittal plane angle between the pelvis position in the erect standing posture and its position at the end of forward trunk bending, as in the FTF measurement.
Straight Leg Raise (SLR) angle | Before and immediately after the intervention
  The SLR angle will be evaluated at baseline and immediately after the intervention. The mean value of the two measurements taken before the intervention will be compared with the mean value of two measurements taken immediately after the intervention. The change in SLR angle values of the less flexible lower limb, expressed as a percentage relative to the initial value, will be used to compare the effect between the PS and PAS groups.
  The rater will raise the participant's lower limb with the knee fully extended until the first sensation of stretch or pain is felt. The angle will then be recorded using the EasyAngle® digital inclinometer, which will be secured with a Velcro strap to the lateral side of the lower limb at the level of the tibial tuberosity.
Hamstring stiffness | Before and immediately after the intervention
  Hamstring stiffness during the SLR maneuver will be measured at baseline and immediately after the intervention. The mean value of the two measurements taken before the intervention will be compared with the mean value of two measurements taken immediately after the intervention. The change in hamstring stiffness of the less flexible lower limb, expressed as a percentage relative to the initial value, will be used to compare the effect between the PS and PAS groups.
  The pulling force applied during the SLR maneuver will be recorded in Newtons using the EasyForce® digital dynamometer.
Pain Visual Analogue Scale (VAS) | Before and immediately after intervention
  Pain will be assessed using the Visual Analogue Scale (VAS), where 0 represents no pain and 100 represents the maximum imaginable pain, at the end of the SLR angle before the intervention. The post-intervention assessment will be recorded at the initial SLR angle or, if the range decreases, at the new end of the SLR angle.
Tampa Scale of Kinesiophobia (TSK-17) | At baseline
  The Tampa Scale of Kinesiophobia (TSK-17) questionnaire will be used to assess fear of movement (kinesiophobia) at baseline. This questionnaire is commonly used for patients with chronic low back pain and demonstrates good psychometric properties. The TSK-17 score ranges from 17 to 68, with higher scores indicating worse outcomes (greater fear of movement) and lower scores indicating better outcomes (less fear of movement).
Score of perceived harmfulness of the movements | At baseline
  Participants will complete a questionnaire assessing their perceived harmfulness of the movements presented in the videos, using a numerical scale (0 - Not harmful at all, 100 - Extremely harmful). A total of seven movements, corresponding to the AKE, SLR, FTF measurements, passive stretching, and three active stretching exercises, will be presented in the videos. The total score and individual scores for each movement will be analyzed.
Skin conductance | During pre-intervention evaluation and during intervention.
  Skin conductance will be measured using a NeuLog device, placed on the fingers of the participant's dominant hand. Fear-related sweat production increases skin conductance and can thus objectively indicate the participant's emotional state.
  The average amplitude of the Skin Conductance Response will be recorded during both the pre-intervention evaluation and the intervention, measured in µS.
Perceived change in flexibility. | Immediately after the intervention
  The participant's declaration of the perceived change in flexibility immediately after the intervention on the movements assessed (AKE, SLR, FTF) will be recorded. The following question will be asked: 'Do you feel a gain in flexibility?' The participant will choose from the following responses: 'No, I feel less flexible,' 'No, I feel no difference,' 'Yes, I feel a little more flexible,' or 'Yes, I feel much more flexible'.

CONTACTS AND LOCATIONS:
Overall Officials: Lech DOBIJA, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - Clermont Ferrand Univbersity HOspital, Louise Michel site, Cébazat, France
  - CHU de Clermont-Ferrand, Clermont-Ferrand

IPD SHARING:
Plan to Share IPD: Yes
The anonymised individual participant data (IPD) will be sheared on demande.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD will be shared on demand, starting from the publication of the primary study results, for up to 10 years after study completion.
Access Criteria: The anonymized IPD will be sent on demand to qualified researchers or institutions.